CLINICAL TRIAL: NCT05095350
Title: Effect of Probiotics on Grade 1 Primary Hypertension and Prehypertension and the Underlying Mechanism: a Randomized Controlled Trial
Brief Title: Effect of Probiotics on Primary Hypertension
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Beijing Municipal Education Commission (Unknown)
Responsible Party: Principal Investigator, Jun Cai, Professor, Director of Hypertension Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROB(2017-BJJW)
Record Dates: First submitted 2021-10-04; First posted 2021-10-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
Keywords: Hypertension; Microbiome; Probiotics; Treatment
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic powder (Experimental): The probiotic powder contains 10 strains from Lactobacillus and Bifidobacterium genus. Participants will orally take two sachets daily and last for 8 weeks.
  Interventions: Biological: Probiotic powder
- Placebo powder (Placebo Comparator): The placebo powder consists of maltodextrin and contains no probiotics. Participants will orally take two sachets daily and last for 8 weeks.
  Interventions: Biological: Placebo powder

INTERVENTIONS:
Biological: Probiotic powder — Probiotic powder containing 10 strains from Lactobacillus and Bifidobacterium genus.
  Arms: Probiotic powder
Biological: Placebo powder — Placebo powder containing maltodextrin and no probiotics.
  Arms: Placebo powder

SUMMARY:
Gut microbiota was found to play a causal role in the pathogenesis of hypertension. Probiotics were shown to have a potential anti-hypertensive effect in human/rodent studies. This study aims to explore the effect, safety, and underlying mechanisms of the combination of probiotics, containing 10 strains from Lactobacillus and Bifidobacterium, on hypertension, compared with placebo.

DETAILED DESCRIPTION:
Background: Primary hypertension is the leading risk factor of cardiovascular diseases and all-cause mortality, and contributes to severe global health burden. Emerging evidence has shown a close association between gut microbiota and hypertension. Fecal transplantation from hypertensive patients/animals to germ-free mice caused elevation of blood pressure, indicating a causal role of gut dysbiosis in hypertension. Probiotics were found to have a potential anti-hypertensive effect in both human and rodent studies. Based on the investigators' previous findings of metagenomics analysis of hypertensive, prehypertensive patients and healthy control, hypertensive and prehypertensive patients were lack of probiotics. Therefore, the investigators developed this study to explore the effect, safety, and underlying mechanisms of the combination of probiotics, containing 10 strains from Lactobacillus and Bifidobacterium, on hypertension, compared with placebo.

Objective: To explore the effect, safety, and underlying mechanisms of the combination of probiotics on grade 1 primary hypertension and prehypertension.

Study Design: A multicenter, randomized, double-blinded, placebo-controlled pilot study.

Data quality control and statistical analysis: The investigators have invited professional statistic analysts to assist in analyzing data and a third party to supervise data quality.

Ethics: The Ethics Committee of Fuwai Hospital approved this study. Informed consent before patient enrollment is required.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~60 years.
2. Grade 1 hypertension and part of prehypertension (initial diagnosis or free from antihypertensive drugs within 2 weeks): 130 mmHg ≤ Average office SBP < 160 mmHg, and/or 85 mmHg ≤ Average office DBP < 100 mmHg, according to the "2018 Chinese Guidelines for Prevention and Treatment of Hypertension" and "National guideline for hypertension management in China (2019)".
3. Patients with informed consent after thorough explanation.

Exclusion Criteria:

1. Antibiotics or probiotics usage within the last 2 weeks.
2. Participants of other clinical trials currently or within last 3 months.
3. Antihypertensive medications usage currently or within last 2 weeks.
4. Diagnosed secondary hypertension
5. History of diabetes mellitus.
6. History of peripheral atherosclerosis.
7. Severe hepatic or renal diseases (ALT >3 times the upper limit of normal value, or end-stage renal disease on dialysis or eGFR <30 mL/min/1.73 m2, or serum creatinine >2.5 mg/dl [>221 μmol/L]).
8. History of stroke (not including lacunar infarction and transient ischemic attack [TIA]).
9. History of coronary heart disease.
10. Sustained atrial fibrillation or arrhythmias at recruitment disturbing the electronic BP measurement.
11. NYHA class III-IV heart failure; Hospitalization for chronic heart failure exacerbation within last 6 months.
12. Severe valvular diseases; Potential for surgery or percutaneous valve replacement within the study period.
13. Dilated cardiomyopathy; Hypertrophic cardiomyopathy; Rheumatic heart disease; Congenital heart disease.
14. Other severe diseases influencing the entry or survival of participants, such as malignant tumor or acquired immune deficiency syndrome.
15. Cognitive impairment or severe neuropsychiatric comorbidities who are incapable of providing their own informed consent.
16. Participants preparing for or under pregnancy and/or lactation.
17. With special diet habits, such as vegetarians.
18. Active gastritis or enteritis; gastrointestinal ulcers or bleeding; post-gastrointestinal surgery, such as intestinal excision.
19. Other conditions inappropriate for recruitment according to the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Change in Office Systolic Blood Pressure (SBP) | From baseline to day 56
  Change in Office Systolic Blood Pressure (SBP)

SECONDARY OUTCOMES:
Change in Office SBP | Baseline, Day28, Day 56, Day 84
  Change in Office SBP
Change in Office Diastolic Blood Pressure (DBP) | Baseline, Day28, Day 56, Day 84
  Change in Office Diastolic Blood Pressure (DBP)
Change in average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Day28, Day 56, Day 84
  Change in average SBP via 24-hour Ambulatory BP Monitoring
Change in average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Day28, Day 56, Day 84
  Change in average DBP via 24-hour Ambulatory BP Monitoring
Change in daytime average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Day28, Day 56, Day 84
  Change in daytime average SBP via 24-hour Ambulatory BP Monitoring
Change in daytime average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Day28, Day 56, Day 84
  Change in daytime average DBP via 24-hour Ambulatory BP Monitoring
Change in nightime average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Day28, Day 56, Day 84
  Change in nightime average SBP via 24-hour Ambulatory BP Monitoring
Change in nightime average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Day28, Day 56, Day 84
  Change in nightime average DBP via 24-hour Ambulatory BP Monitoring
Number of Participants with Adverse Events (AEs) as a Measure of Safety | Baseline, Day28, Day 56, Day 84
  Number of Participants with Adverse Events (AEs) as a Measure of Safety
Changes in Intestinal Microbiota Composition Pre- and Post-intervention via Metagenomic Analysis | Baseline, Day28, Day 56, Day 84
  Intestinal microbiota composition is obtained through sequencing of DNAs from feces samples and bioinformatic analysis. Changes in the intestinal microbiota composition before and after intervention (probiotics or placebo) is defined as a secondary outcome. This is stratified by: 1. Randomization (probiotics or placebo); 2. Changes in office SBP.
Changes in Intestinal Microbiota Function Pre- and Post-intervention via Metagenomic Analysis | Baseline, Day28, Day 56, Day 84
  Intestinal microbiota function is obtained through sequencing of DNAs from feces samples and bioinformatic analysis according to functions related to detected genes. Changes in the intestinal microbiota function before and after intervention (probiotics or placebo) is defined as a secondary outcome. This is stratified by: 1. Randomization (probiotics or placebo); 2. Changes in office SBP.
Changes in Intestinal Metabolite Composition Pre- and Post-intervention via Metabolomic Analysis | Baseline, Day28, Day 56, Day 84
  Metabolomics analysis is a quantitative analysis of all metabolites in the sample. Metabolites in feces are detected using liquid or gas chromatography combined with mass spectrometry, and the composition and abundance of each metabolite are obtained. Changes in the intestinal metabolite composition before and after intervention (probiotics or placebo) is defined as a secondary outcome. This is stratified by: 1. Randomization (probiotics or placebo); 2. Changes in office SBP.
  Randomisation Change in Office SBP
Changes in Serum Metabolite Composition Pre- and Post-intervention via Metabolomic Analysis | Baseline, Day28, Day 56, Day 84
  Metabolomics analysis is a quantitative analysis of all metabolites in the sample. Metabolites in serum are detected using liquid or gas chromatography combined with mass spectrometry, and the composition and abundance of each metabolite are obtained. Changes in the serum metabolite composition before and after intervention (probiotics or placebo) is defined as a secondary outcome. This is stratified by: 1. Randomization (probiotics or placebo); 2. Changes in office SBP.
  Randomisation Change in Office SBP
Change in Fasting Blood Glucose Level | Baseline, Day 56
  Change in Fasting Blood Glucose Level
Change in Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol) | Baseline, Day 56
  Change in Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol)
Change in Blood Uric Acid | Baseline, Day 56
  Change in Blood Uric Acid
Change in Body Mass Index | Baseline, Day 56
  Change in Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: JUN CAI, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (6):
- China (6):
  - Fu Wai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Longgang District People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Affiliated Hospital of Baotou Medical Collage, Baotou, Neimenggu
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

REFERENCES:
- [Background] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Background] Wilck N, Matus MG, Kearney SM, Olesen SW, Forslund K, Bartolomaeus H, Haase S, Mahler A, Balogh A, Marko L, Vvedenskaya O, Kleiner FH, Tsvetkov D, Klug L, Costea PI, Sunagawa S, Maier L, Rakova N, Schatz V, Neubert P, Fratzer C, Krannich A, Gollasch M, Grohme DA, Corte-Real BF, Gerlach RG, Basic M, Typas A, Wu C, Titze JM, Jantsch J, Boschmann M, Dechend R, Kleinewietfeld M, Kempa S, Bork P, Linker RA, Alm EJ, Muller DN. Salt-responsive gut commensal modulates TH17 axis and disease. Nature. 2017 Nov 30;551(7682):585-589. doi: 10.1038/nature24628. Epub 2017 Nov 15. PMID 29143823
- [Background] Robles-Vera I, Toral M, de la Visitacion N, Sanchez M, Gomez-Guzman M, Romero M, Yang T, Izquierdo-Garcia JL, Jimenez R, Ruiz-Cabello J, Guerra-Hernandez E, Raizada MK, Perez-Vizcaino F, Duarte J. Probiotics Prevent Dysbiosis and the Rise in Blood Pressure in Genetic Hypertension: Role of Short-Chain Fatty Acids. Mol Nutr Food Res. 2020 Mar;64(6):e1900616. doi: 10.1002/mnfr.201900616. Epub 2020 Feb 6. PMID 31953983
- [Background] Khalesi S, Sun J, Buys N, Jayasinghe R. Effect of probiotics on blood pressure: a systematic review and meta-analysis of randomized, controlled trials. Hypertension. 2014 Oct;64(4):897-903. doi: 10.1161/HYPERTENSIONAHA.114.03469. Epub 2014 Jul 21. PMID 25047574